CLINICAL TRIAL: NCT00038220
Title: A Phase I/II, Open Label Study to Evaluate the Ability of Combination Therapy With ABT-378/Ritonavir (Kaletra), Lamivudine (Epivir), Efavirenz (Sustiva)and Tenofovir DF to Completely Suppress Viral Replication in Subjects Infected With HIV-1
Brief Title: Effectiveness of ABT-378/Ritonavir Plus Lamivudine Plus Efavirenz Plus Tenofovir DF in HIV-Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M00-154; NCT00006189 (obsolete NCT alias)
Record Dates: First submitted 2002-05-29; First posted 2002-05-30 (Estimated); Last update posted 2006-07-27 (Estimated); Status verified 2006-07

CONDITIONS: HIV Infections
Keywords: HIV
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir; efavirenz; Lamivudine; Tenofovir

INTERVENTIONS:
Drug: Lopinavir/ritonavir
Drug: Efavirenz
Drug: Lamivudine
Drug: Tenofovir DF

SUMMARY:
The purpose of this study is to see if a novel 4-drug anti-HIV combination can suppress the growth of HIV in patients infected with the virus.

ELIGIBILITY:
Inclusion Criteria:

* Have HIV Infection.
* Age 18 to 65 years old.
* Show no signs of recent illness other than HIV infection.
* Agree to use a barrier method of birth control during the study and for 30 days after study.

Exclusion Criteria:

* Are unable to follow study requirements (in the opinion of the investigator).
* Are pregnant or breast-feeding.
* Are unable to take medications by mouth.
* Have chronic nausea or vomiting.
* Have cancer other than Kaposi's sarcoma or basal cell carcinoma.
* Have active, serious infections (other than HIV) requiring antibiotic injections within 15 days prior to screening.
* Are taking any medications that are not allowed with ABT-378/r and efavirenz.
* Are taking or have taken any other experimental drugs, antiretroviral drugs, or drugs that affect the immune system within 30 days of start of study without consent of the medical monitor.
* Are receiving or have received radiation therapy within 30 days of start of study without consent of the medical monitor.
* Have a history of drug abuse or mental illness that would prevent the patient from following the protocol requirements.
* Have a history of kidney or bone disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2000-07

PRIMARY OUTCOMES:
Proportion of subjects in each group demonstrating complete suppression of viral replication at Week 144.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Brun, M.D., Study Director — Head, Antiviral Global Project Team
Locations (1):
- Aaron Diamond AIDS Research Center - Rockefeller University, New York, New York, United States